CLINICAL TRIAL: NCT04738461
Title: The Effectiveness of Telerehabilitation in Patients With Subacromial Pain Syndrome: a Randomized Controlled Trial
Brief Title: The Effectiveness of Telerehabilitation in Patients With Subacromial Pain Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: postponed to a later date
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BI280121
Record Dates: First submitted 2021-01-31; First posted 2021-02-04 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Subacromial Pain Syndrome
Keywords: Subacromial Pain Syndrome; Subacromial ImpingementSyndrome; telerehabilitation; physiotherapy
MeSH Terms: interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: Prospective, triple-blinding, randomized controlled and 3-arm parallel group design clinical study. 3 arms of the study were planned to consist of telerehabilitation group, standard physiotherapy group and home exercise group.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will not be able to be blinded due the inherent of interventions. Staff members who are responsible for statistical analysis, investigators and outcome assessors will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Telerehabilitation (Experimental): Telerehabilitation program will be applied 5 days a week for 3 weeks to patients in the telerehabilitation group. A physiatrist will meet with patients via videoconferencing over the internet and guide the program.
  Interventions: Other: Telerehabilitation
- Standard Physiotherapy (Active Comparator): Patients in the standard physiotherapy group will receive one-to-one physiotherapy sessions in the hospital 5 days a week for 3 weeks. In these sessions, active-passive exercises accompanied by a physiotherapist and physical therapy methods (electrotherapy and thermotherapy) will be applied in accordance with the standard procedure according to the patient's needs.
  Interventions: Other: Standard Physiotherapy
- Home exercise group (Active Comparator): The home exercise program was explained to the patients in the control group by the physiotherapist and the relevant brochures were delivered to the patients. Home exercise program will consist of telerehabilitation group exercises. However, patients will be not under any supervision and exercise themselves at home.
  Interventions: Other: Home Exercise Group

INTERVENTIONS:
Other: Telerehabilitation — The Posterior Glenohumeral Capsule Stretching Exercise, Pectoral Stretching Exercise, Push-up Against Wall Exercise, Scapular Plan Exercise, 90 Degree Shoulder Flexion Exercise, Isometric External Rotation Exercise and Isometric Internal Rotation Exercise will be applied according to the severity of the disease and the size of the disability.
  Arms: Telerehabilitation
Other: Standard Physiotherapy — Active-passive exercises accompanied by a physiotherapist and physical therapy methods (electrotherapy and thermotherapy) will be applied in accordance with the standard procedure according to the patient's needs.
  Arms: Standard Physiotherapy
Other: Home Exercise Group — The same exercise program applied to telerehabilitation group.
  Arms: Home exercise group

SUMMARY:
The main hypothesis of the study is that telerehabilitation is an effective treatment method and it is not inferior than standard physiotherapy.The aim of this study is to evaluate the effectiveness of telerehabilitation in patients with subacromial pain syndrome by comparing it with standard physiotherapy.

DETAILED DESCRIPTION:
Subacromial pain syndrome formerly known as subacromial impingement syndrome is the cause of approximately 44% to 65% of pain complaints related to the shoulder. Methods such as immobilization, drug therapy, injection techniques, physical therapy modalities and therapeutic exercises, manual therapy, acupuncture and surgery can be used in the treatment of the disease. Due to the Coronavirus disease 2019 (COVID-19) pandemic that started in Wuhan province of China in December 2019, the problems in patients' access to hospitals and rehabilitation services caused telerehabilitation to be on the agenda. Telerehabilitation can be summarized as the delivery of rehabilitation services to those in need by using communication technologies. This method covers the steps of evaluation, monitoring, prevention, intervention, control, training, and consultation. Although there are many studies on the effectiveness of telerehabilitation in the literature, there is no study on the superiority of telerehabilitation, physical therapy under supervision and home exercise program over each other.

ELIGIBILITY:
Inclusion Criteria:

* Having subacromial pain for at least 2 weeks
* Positive result of Hawkins-Kennedy, painful arc or infraspinatus muscle strength tests .
* To have internet access and equipment to participate in videoconference .
* Being literate and not having cognitive dysfunction.

Exclusion Criteria:

* Positive drop arm test
* Signs of adhesive capsulitis (restriction in range of motion-especially in abduction and external rotation)
* Grade 3 or full thickness rotator cuff tear
* Labral tears and other intraarticular structural pathologies
* History of shoulder surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Pain Intensity at 1 and 3 months | Baseline, one and three month after the randomisation
  Patients will be asked to mark their pain by giving a score between zero (no pain) and 10 (the most severe pain) on a 10 cm long visual analog scale (VAS) during each visits.

SECONDARY OUTCOMES:
Change from Baseline SPADI total score at 1 and 3 months | Baseline, one and three month after the randomisation
  The Shoulder Pain and Disability Index (SPADI) is a questionnaire with a total of 13 questions developed to measure shoulder pain and associated disability. In the subgroup of the pain, the patient is asked to express the severity of him/her pain by giving a score between zero (no pain) and 10 (the most severe pain) during different activities in the last week. In the subgroup of disability, the patient is asked to score between zero (no difficulty) and 10 (receiving assistance) how hard they have experienced during different activities in the last week. Zero points indicate maximum well-being, 130 points indicate maximum disability.

OTHER OUTCOMES:
Change from baseline range of motion of shoulder at 1 and 3 months | Baseline, one and three month after the randomisation
  Range of motion of the Shoulder will be evaluated with a standard goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Bugra Ince, MD, Principal Investigator — Bezmialem Vakif University; Mustafa Huseyin Temel, MD, Principal Investigator — Uskudar State Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Cam and Sakura City Hospital, Istanbul
  - Medipol Mega University Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No
Data sharing will be done on request

REFERENCES:
- [Background] Garving C, Jakob S, Bauer I, Nadjar R, Brunner UH. Impingement Syndrome of the Shoulder. Dtsch Arztebl Int. 2017 Nov 10;114(45):765-776. doi: 10.3238/arztebl.2017.0765. PMID 29202926
- [Background] Carbonaro N, Lucchesi I, Lorusssi F, Tognetti A. Tele-monitoring and tele-rehabilitation of the shoulder muscular-skeletal diseases through wearable systems. Annu Int Conf IEEE Eng Med Biol Soc. 2018 Jul;2018:4410-4413. doi: 10.1109/EMBC.2018.8513371. PMID 30441330